CLINICAL TRIAL: NCT03019965
Title: Efficacy and Safety of the Administration of Betalactam Antibiotics in Continuous or Extended Infusion Compared to Intermittent Infusion in Patients With Sepsis in Two Pediatric Third-level Care Hospitals
Brief Title: Efficacy of Betalactam Antibiotics in Prolonged Infusion Compared to Intermittent in Pediatric Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); Hospital Infantil de Mexico Federico Gomez (Other); Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Yazmín Del Carmen Fuentes Pacheco, Pediatric Infectious Disease, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-785-099
Record Dates: First submitted 2016-12-26; First posted 2017-01-13 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Tazobactam; Meropenem

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Intermittent Piperacillin/tazobactam (Active Comparator): Piperacillin/tazobactam 300mg/kg/day, divided into 4 doses/day, diluted in 5% glucose solution, at a concentration of 50mg/ml, to be administered in 30 minutes infusion every 6 hours.
  Interventions: Drug: Intermittent Piperacillin/tazobactam
- Continuous Piperacillin/tazobactam (Experimental): Piperacillin/tazobactam initial doses 75mg/kg in 30 minutes infusion, immediately thereafter continue 300mg/kg/day, diluted in 5% glucose solution, at a concentration of 50mg/ml, to be administered in 24 hours infusion every 24 hours, as determined by antibiotic stability at room temperature.
  Interventions: Drug: Continuous Piperacillin/tazobactam
- Intermittent Imipenem (Active Comparator): Imipenem 80mg/kg/day, divided into 4 doses/day, diluted in 0.9% saline solution, at a concentration of 7mg/ml, to be administered in 60 minutes infusion every 6 hours.
  Interventions: Drug: Intermittent Imipenem
- Extended Imipenem (Experimental): Imipenem initial doses 20mg/kg in 60 minutes infusion, immediately thereafter continue 80mg/kg/day, divided into 4 doses/day, diluted in 0.9% saline solution, at a concentration of 7mg/ml, to be administered in 6 hours infusion every 6 hours, as determined by antibiotic stability at room temperature.
  Interventions: Drug: Extended Imipenem
- Intermittent Meropenem (Active Comparator): Meropenem 100mg/kg/day, divided into 3 doses/day, diluted in 0.9% saline solution, at a concentration of 7mg/ml, to be administered in 60 minutes every 8 hours.
  Interventions: Drug: Intermittent Meropenem
- Extended Meropenem (Experimental): Meropenem initial doses 35mg/kg in 60 minutes infusion, immediately thereafter continue 100mg/kg/day, divided into 3 doses/day, diluted in 0.9% saline solution at a concentration of 7mg/ml, to be administered in 8 hours infusion every 8 hours, as determined by antibiotic stability at room temperature.
  Interventions: Drug: Extended Meropenem

INTERVENTIONS:
Drug: Intermittent Piperacillin/tazobactam — Piperacillin/tazobactam administered in 30 minutes infusion.
  Other Names: Intermittent Infusion of Piperacillin/tazobactam; PiSA
  Arms: Intermittent Piperacillin/tazobactam
Drug: Continuous Piperacillin/tazobactam — Piperacillin/tazobactam administered in 24 hours infusion.
  Other Names: Continuous Infusion of Piperacillin/tazobactam; PiSA
  Arms: Continuous Piperacillin/tazobactam
Drug: Intermittent Imipenem — Imipenem administered in 60 minutes infusion.
  Other Names: Intermittent Infusion of Imipenem; PiSA
  Arms: Intermittent Imipenem
Drug: Extended Imipenem — Imipenem administered in 6 hours infusion.
  Other Names: Extended Infusion of Imipenem; PiSA
  Arms: Extended Imipenem
Drug: Intermittent Meropenem — Meropenem administered in 60 minutes infusion.
  Other Names: Intermittent Infusion of Meropenem; Kener; Merrem, AstraZeneca
  Arms: Intermittent Meropenem
Drug: Extended Meropenem — Meropenem administered in 8 hours infusion.
  Other Names: Extended Infusion of Meropenem; Kener; Merrem, AstraZeneca
  Arms: Extended Meropenem

SUMMARY:
This study evaluates the efficacy and safety of the administration of betalactam antibiotics in prolonged infusion compared to intermittent infusion in children with sepsis. Half of participants will receive piperacillin/tazobactam, imipenem or meropenem in continuous or extended infusion, while the other half will receive piperacillin/tazobactam, imipenem or meropenem in intermittent infusion.

DETAILED DESCRIPTION:
Sepsis is the leading cause of morbidity and mortality in hospitalised patients globally. Betalactams are time-dependent antibiotics, and so, the duration of time for which the free drug plasma concentration remains above the minimum inhibitory concentration (fT > MIC) is the pharmacokinetic/pharmacodynamic index associated with bacterial killing and clinical improvement. Numerous studies have demonstrated that continuous infusion (infusion in 24 hours) and extended infusion (through prolonging the infusion time to greater than 3 hours) allows the maintenance of concentrations above the MIC for a longer period of time within the dosing interval (30 minute or 1 hour), and so, capitalises on the pharmacodynamic properties of betalactams and maximises bacterial killing, therefore potentially improving clinical outcomes. In adult patients, the several studies suggest that prolonged infusion may offer clinical benefits and significant reduction in mortality without increasing the risk of toxicity, however, there is limited information about these dosing strategies in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sepsis, who have been evaluated by an infectious physician and are candidates to receive piperacillin/tazobactam, imipenem or meropenem as empiric treatment.

Exclusion Criteria:

* Patients with a history of allergy to one or more of the proposed antibiotics.
* Patients with chronic kidney disease or acute renal failure.
* Patients with acute liver failure of any cause.
* Patients in palliative or supportive care only.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 426 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yazmín del Carmen Fuentes, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (2):
- Mexico (2):
  - Hospital Infantil de México Federico Gómez, Mexico City, Mexico City
  - Instituto Mexicano del Seguro Social, Mexico City, Mexico City

IPD SHARING:
Plan to Share IPD: No
Identified individual participant data for all primary and secondary outcome measures will be made available within six months of study completion

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: the pre-specified intent was to only compare "Intermittent" and "Prolonged" Arm/Groups with the grouping of betalactam antibiotics (imipenem, meropenem and piperacillin/tazobactam)
Groups:
- Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem: Piperacillin/tazobactam 300mg/kg/day, divided into 4 doses/day, diluted in 5% glucose solution, at a concentration of 50mg/ml, to be administered in 30 minutes infusion every 6 hours.
  Intermittent Piperacillin/tazobactam: Piperacillin/tazobactam administered in 30 minutes infusion.
  Imipenem 80mg/kg/day, divided into 4 doses/day, diluted in 0.9% saline solution, at a concentration of 7mg/ml, to be administered in 60 minutes infusion every 6 hours.
  Intermittent Imipenem: Imipenem administered in 60 minutes infusion. Meropenem 100mg/kg/day, divided into 3 doses/day, diluted in 0.9% saline solution, at a concentration of 7mg/ml, to be administered in 60 minutes every 8 hours.
  Intermittent Meropenem: Meropenem administered in 60 minutes infusion.
- Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem: Piperacillin/tazobactam initial doses 75mg/kg in 30 minutes infusion, immediately thereafter continue 300mg/kg/day, diluted in 5% glucose solution, at a concentration of 50mg/ml, to be administered in 24 hours infusion every 24 hours, as determined by antibiotic stability at room temperature.
  Continuous Piperacillin/tazobactam: Piperacillin/tazobactam administered in 24 hours infusion.
  Imipenem initial doses 20mg/kg in 60 minutes infusion, immediately thereafter continue 80mg/kg/day, divided into 4 doses/day, diluted in 0.9% saline solution, at a concentration of 7mg/ml, to be administered in 6 hours infusion every 6 hours, as determined by antibiotic stability at room temperature.
  Extended Imipenem: Imipenem administered in 6 hours infusion.
  Meropenem initial doses 35mg/kg in 60 minutes infusion, immediately thereafter continue 100mg/kg/day, divided into 3 doses/day, diluted in 0.9% saline solution at a concentration of 7mg/ml, to be administered in 8 hours infusion every 8 hours, as determined by antibiotic stability at room temperature.
  Extended Meropenem: Meropenem administered in 8 hours infusion.
Period: Overall Study
Arm/Group | Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem | Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem
Started | 211 | 215
Completed | 201 | 202
Not Completed | 10 | 13
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — viral or fungal infection | 3 | 4
Not completed — acute liver failure in the first 24 hours of randomization | 4 | 5
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem | Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem | Total
Number analyzed (Participants) | 201 | 202 | 403
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 201 | 202 | 403
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 6 [0 to 17] | 6 [0 to 17] | 6 [0 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 91 | 182
  Male | 110 | 111 | 221
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 201 | 202 | 403
Comorbidity [Count of Participants; unit: Participants] | 196 | 187 | 383
Comorbid conditions [Count of Participants; unit: Participants] — Population: Comorbidity only was in 196 patients in intermittent infusion group and 187 patients in prolonged infusion group.
  Participants
    number analyzed (Participants) | 196 | 187 | 383
    Neoplastic | 125 | 133 | 258
    Gastrointestinal | 20 | 15 | 35
    Neurological | 8 | 11 | 19
    Neonatal | 2 | 3 | 5
    Cardiovascular | 15 | 8 | 23
    Respiratory | 2 | 2 | 4
    Hematologic/immunologic | 11 | 4 | 15
    Metabolic | 1 | 1 | 2
    Renal | 1 | 0 | 1
    Genetic | 11 | 9 | 20
    Stem cell transplant | 0 | 1 | 1
Hospital stay prior to enrollment to the study protocol [Count of Participants; unit: Participants] — number of participants who had been hospitalized for at least 24 hours prior to enrollment to the study protocol
  Participants | 113 | 122 | 235
septic shock at enrollment [Count of Participants; unit: Participants] | 49 | 61 | 110
B-lactam antibiotic [Count of Participants; unit: Participants]
  piperacillin/tazobactam | 109 | 108 | 217
  imipenem | 39 | 42 | 81
  meropenem | 53 | 52 | 105
type of infection [Count of Participants; unit: Participants]
  febrile neutropenia | 69 | 55 | 124
  intraabdominal | 40 | 55 | 95
  respiratory tract | 34 | 27 | 61
  bacteremia | 30 | 35 | 65
  skin and soft tissue | 11 | 10 | 21
  unknown | 11 | 14 | 25
  urinary tract | 6 | 6 | 12
Number of participants with organisms identified [Count of Participants; unit: Participants] | 75 | 86 | 161

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response
Description: Resolution. Disappearance of all signs and symptoms related to the infection.
  Failure. Insufficient lessening of the signs and symptoms of infection to qualify as improvement, including death or indeterminate (no evaluation possible, for any reason).
Time Frame: Number of participants with clinical response at 14 days after antibiotic cessation, up to an average of 28 days or the day of your discharge if this occurred before 14 days after antibiotic cessation.
Population: The efficacy of the maneuver was evaluated by frequency of clinical response and calculation of the absolute risk reduction and the number needed to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem | Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem
Number analyzed (Participants) | 201 | 202
Participants | 178 | 169
Statistical Analysis 1: Comparison: Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem vs Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem; Test type: Superiority; p = 0.156, Chi-squared; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.87 to 1.02]; The efficacy of the maneuver was evaluated by calculating the absolute risk reduction and the number needed to treat

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Any harmful, undesirable, potentially serious and life threatening effects occurring during or after administration of the antibiotics proposed in this study (piperacillin / tazobactam, imipenem or meropenem), was evaluated as: none or adverse event classified according to the intensity of the clinical manifestation (severity) as: mild, moderate or severe and for each antibiotic.
Time Frame: Number of participants with adverse events evaluated by an physician at the time of administration of antibiotics, up to an average to 24 hours after the study drug cessation.
Population: evaluation of the safety of the intervention with analysis of the frequency of adverse events by treatment group
Measure: Count of Participants; unit: Participants
Arm/Group | Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem | Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem
Number analyzed (Participants) | 201 | 202
Participants | 1 | 3
Statistical Analysis 1: Comparison: Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem vs Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem; Test type: Superiority; p = 0.722, Chi-squared; Risk Ratio (RR) = 2.98, 95% CI 2-sided [0.31 to 28.45]

ADVERSE EVENTS:
Time Frame: adverse events by the mode of administration: intermittent or prolonged, evaluated during the time of administration, up to an average 24 hours after administration of the antibiotics proposed.
Description: pre-specified intent was to only compare "Intermittent" and "Prolonged" Arm/Groups with the grouping of antibiotics betalactam (imipenem, meropenem and piperacillin/tazobactam)
Arm/Group | Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem | Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem
All-Cause Mortality (participants affected / at risk) | 17/201 | 19/202
Serious Adverse Events (participants affected / at risk) | 0/201 | 0/202
Other Adverse Events (participants affected / at risk) | 1/201 | 3/202
OTHER ADVERSE EVENTS (reported when occurring in more than 1.49% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent. Piperacillin/Tazobactam, Imipenem, Meropenem (N=201) | Prolonged Infusion. Continuous Piperacillin/Tazobactam, Extended Imipenem, Extended Meropenem (N=202)
moderate adverse event (Gastrointestinal disorders) | 1 (1) | 3 (3) — vomiting, diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT03019965/Prot_SAP_000.pdf